CLINICAL TRIAL: NCT04610203
Title: Glycaemic, Insulinaemic, Gastric Inhibitory Polypeptide (GIP) and Glucagon-like Peptide-1 (GLP-1) Response for Glucose, Glucose With 25 g Nutralys S85 Plus and Glucose With 50 g Nutralys S85 Plus
Brief Title: Glycaemic Response, Insulinaemic Response, GLP-1 and GIP Testing of Food Product Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: Roquette Freres (Industry)
Responsible Party: Principal Investigator, Dr. Sangeetha Thondre, Principal Investigator, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CPS 18-439; pfact 9806 (Other: Oxford Brookes University)
Record Dates: First submitted 2020-10-10; First posted 2020-10-30 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Healthy
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: randomised, repeat measure, crossover design trial
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucose (Placebo Comparator): Glucose - 50 g
  Interventions: Dietary Supplement: 50 g Glucose
- Nutralys S85 Plus 25 g (Experimental): Nutralys S85 Plus Pea Protein 25 g + 50 g Glucose
  Interventions: Dietary Supplement: 25 g Nutralys Pea Protein
- Nutralys S85 Plus 50 g (Experimental): Nutralys S85 Plus Pea Protein 50 g + 50 g Glucose
  Interventions: Dietary Supplement: 50 g Nutralys S85 Plus.

INTERVENTIONS:
Dietary Supplement: 25 g Nutralys Pea Protein — To determine the glycaemic response, insulinaemic response, GIP response and GLP-1 response to 50g Glucose +25g Nutralys S85 Plus
  Arms: Nutralys S85 Plus 25 g
Dietary Supplement: 50 g Nutralys S85 Plus. — To determine the glycaemic response, insulinaemic response, GIP response and GLP-1 response to 50g Glucose+50 g Nutralys S85 Plus .
  Arms: Nutralys S85 Plus 50 g
Dietary Supplement: 50 g Glucose — To determine the glycaemic response, insulinaemic response, GIP response and GLP-1 response to 50g Glucose
  Arms: Glucose

SUMMARY:
The aim of this study was to compare the glycaemic response, insulinaemic response, GIP response and GLP-1 response to glucose, 25 g Nutralys S85 Plus and 50 g Nutralys S85 Plus using a single-blind, randomised, repeat measure, crossover design trial.

DETAILED DESCRIPTION:
The aims of this study were to examine:

* Phase I - the glycaemic response (GR) and insulinaemic response (IR) to:

  * 50 g available carbohydrate
  * 50 g available carbohydrate + protein (dose 1)
  * 50 g available carbohydrate + protein (dose 2)
* Phase II - the GLP-1 and GIP response to:

  * 50 g available carbohydrate
  * 50 g available carbohydrate + protein (dose 1)
  * 50 g available carbohydrate + protein (dose 2)

A single-blind, randomised, repeat measure, crossover design trial was used to study the response following consumption of three meals: one reference meal (50 g available carbohydrate) and two test meals (50 g available carbohydrate with protein dose 1 and 50 g available carbohydrate with protein dose 2). The study was conducted in two phases:

* Phase I: glycaemic response (GR), insulinaemic response (IR)
* Phase II: GLP-1 response and GIP response

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years
* Body mass index (BMI) less than 30kg/m2

Exclusion Criteria:

* Pregnant or lactating
* Fasting blood glucose value > 6.1 mmol/l
* Any known food allergy or intolerance
* Medical condition(s) or medication(s) known to affect glucose regulation or appetite and/or which influence digestion and absorption of nutrients
* Known history of diabetes mellitus or the use of antihyperglycaemic drugs or insulin to treat diabetes and related conditions
* Major medical or surgical event requiring hospitalization within the preceding 3 months
* Use of steroids, protease inhibitors or antipsychotics (all of which have major effects on glucose metabolism and body fat distribution).
* Unable to comply with experimental procedures or did not follow GR testing safety guidelines.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose response from baseline for 3 hours | 3 hours
  Change in postprandial blood glucose response from baseline was measured at 15 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours
Change in plasma insulin response from baseline for 3 hours | 3 hours
  Change in postprandial plasma insulin response from baseline was measured at 15 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours
Area under the blood glucose concentration versus time curve | 3 hours
  Area under the blood glucose concentration versus time curve was calculated by trapezoidal rule
Area under the plasma insulin concentration versus time curve | 3 hours
  Area under the plasma insulin concentration versus time curve was calculated by trapezoidal rule
Peak blood glucose concentration (Cmax) | 0-3 hours
  Peak blood glucose concentration (Cmax) after consumption of the test food
Peak plasma insulin concentration (Cmax) | 0-3 hours
  Peak plasma insulin concentration (Cmax) after consumption of the test food
Time of blood glucose peak (Tmax) | 0-3 hours
  Time of blood glucose peak after consumption of the test food
Time of plasma insulin peak (Tmax) | 0-3 hours
  Time of plasma insulin peak after consumption of the test food

SECONDARY OUTCOMES:
Change in GLP-1 from baseline for 3 hours | 3 hours
  Change in GLP-1 from baseline was measured at 15 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours
Change in GIP from baseline for 3 hours | 3 hours
  Change in GIP from baseline was measured at 15 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours
Area under the plasma GLP-1 concentration versus time curve | 3 hours
  Area under the plasma GLP-1 concentration versus time curve was calculated by trapezoidal rule
Area under the plasma GIP concentration versus time curve | 3 hours
  Area under the plasma GIP concentration versus time curve was calculated by trapezoidal rule
Peak plasma GLP-1 concentration (Cmax) | 0-3 hours
  Peak plasma GLP-1 concentration (Cmax) after consumption of the test food
Peak plasma GIP concentration (Cmax) | 0-3 hours
  Peak plasma GIP concentration (Cmax) after consumption of the test food
Time of plasma GLP-1 peak (Tmax) | 0-3 hours
  Time of plasma GLP-1 peak after consumption of the test food
Time of plasma GIP peak (Tmax) | 0-3 hours
  Time of plasma GIP peak after consumption of the test food

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Thondre, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes Centre for Nutrition and Health, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siahanidou T, Margeli A, Kappis A, Papassotiriou I, Mandyla H. Circulating visfatin levels in healthy preterm infants are independently associated with high-density lipoprotein cholesterol levels and dietary long-chain polyunsaturated fatty acids. Metabolism. 2011 Mar;60(3):389-93. doi: 10.1016/j.metabol.2010.03.002. Epub 2010 Mar 31. PMID 20359723
- See also: 23. Food Products-Determination of the glycaemic index (GI) and recommendation for food classification. — http://www.iso.org/standard/43633.html
- Available data/document: Study Protocol — http://drive.google.com/drive/folders/1H_y4bMle13r4wOG8YyapreznKUFG8cT_
- Available data/document: Informed Consent Form — http://drive.google.com/drive/folders/1H_y4bMle13r4wOG8YyapreznKUFG8cT_
- Available data/document: Clinical Study Report — http://drive.google.com/drive/folders/1H_y4bMle13r4wOG8YyapreznKUFG8cT_
- Available data/document: Individual Participant Data Set — http://drive.google.com/drive/folders/1H_y4bMle13r4wOG8YyapreznKUFG8cT_
- Available data/document: Statistical Analysis Plan — http://drive.google.com/drive/folders/1H_y4bMle13r4wOG8YyapreznKUFG8cT_ — Included in the Study Protocol and Clinical Study report

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04610203/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT04610203/ICF_001.pdf